CLINICAL TRIAL: NCT02199054
Title: Evaluation of Functional Snack Foods Containing Safflower Oil and Soy on Endpoints of Energy Metabolism in Postmenopausal Women With Metabolic Syndrome
Brief Title: Functional Snack Foods With Safflower Oil and Soy in Postmenopausal Women Having Metabolic Syndrome
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Yael Vodovotz, Professor, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 2014H0045; 2013 (Other Grant/Funding Number: Food Innovation Center)
Record Dates: First submitted 2014-07-19; First posted 2014-07-24 (Estimated); Last update posted 2025-02-17 (Actual); Status verified 2024-02

CONDITIONS: Metabolic Syndrome; Overweight
Keywords: Snack Foods; Safflower Oil; Soy; Postmenopausal women; Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome; Overweight

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Run-in Intervention (Placebo Comparator): Control wheat pretzel bites (12 pieces total) will be consumed with a flavored oil dip containing a standardized quantity of triglycerides (50 g long chain fatty acids) at the start of a 7 hour clinic visit as well as 6 pieces of control wheat pretzels will be eaten twice a day (total of 12 pieces/day) for 28 days. During these 28 days, participants will monitor their oil consumption and maintain a legume-free diet.
  Interventions: Other: control wheat pretzels
- Wheat-Safflower Oil Arm (Active Comparator): Wheat-safflower oil pretzel bites (12 pieces total) will be consumed with a flavored oil dip containing a standardized quantity of triglycerides (50 g long chain fatty acids) at the start of a 7 hour clinic visit as well as 6 pieces of wheat-safflower oil pretzels will be eaten twice a day (total of 12 pieces/day) for 28 days. During these 28 days, participants will monitor their oil consumption and maintain a legume-free diet.
  Interventions: Other: wheat-safflower oil pretzels
- Soy-Safflower Oil Arm (Active Comparator): Soy-safflower oil pretzel bites (12 pieces total) will be consumed with a flavored oil dip containing a standardized quantity of triglycerides (50 g long chain fatty acids) at the start of a 7 hour clinic visit as well as 6 pieces of soy-safflower oil pretzels will be eaten twice a day (total of 12 pieces/day) for 28 days. During these 28 days, participants will monitor their oil consumption and maintain a legume-free diet.
  Interventions: Other: soy-safflower oil pretzels

INTERVENTIONS:
Other: wheat-safflower oil pretzels — Each serving (6 pieces) of the wheat-safflower oil pretzel contains 6 grams of safflower oil. Ingredients in the pretzel are high gluten wheat flour, safflower oil, sugar, yeast, salt, and ascorbic acid.
  Arms: Wheat-Safflower Oil Arm
Other: soy-safflower oil pretzels — Each serving (6 pieces) of the soy-safflower oil pretzel contains 6 grams of safflower oil. Ingredients in the pretzel are high gluten wheat flour, soy flour, soymilk, safflower oil, sugar, yeast, salt, and ascorbic acid.
  Arms: Soy-Safflower Oil Arm
Other: control wheat pretzels — Each serving (6 pieces) of the control wheat pretzel contains 6 grams of vegetable shortening. Ingredients in the pretzel are high gluten wheat flour, vegetable shortening, sugar, yeast, salt, and ascorbic acid.
  Arms: Run-in Intervention

SUMMARY:
This research study is being done to help researchers develop new dietary options for menopausal women to maintain a healthy weight by developing more nutritious snacks that have health benefits. From this study, the researchers hope to gain understanding on how menopausal women with metabolic syndrome digest and absorb foods with safflower oil on its own and when combined with soy. The research team hypothesize that the two different types of pretzels may be processed by your body differently and that components in the pretzel snacks may be helpful for preventing diseases like obesity and cancer. Safflower oil and soybeans contain many natural chemicals that may benefit human health. However, this relationship is not well understood. This study will look at the impact of the pretzel snacks on your blood fat and glucose levels as well as a group of chemicals found in soy called "isoflavones". Isoflavones are natural chemicals found commonly in soybeans or foods made from them.

Participants will be screened to determine if they qualify in meeting the study requirements. Participants cannot have a known allergy to dairy, soy, safflower oil, or wheat protein. Also, participants will be asked to stop eating legumes (beans, peas, soy protein, sprouts and peanuts) and to document the oils they eat for the entire 14 weeks of this study. The study will require five visits to the Ohio State University Clinical Research Center (CRC) which part of the Ohio State University's Center for Clinical and Translational Sciences. Once the investigators have determined that you qualify for this study and you decide to participate, you will be consuming three different pretzels each for one month, starting with a control pretzel. After the control pretzel treatment period, you will be randomly assigned (like the "flip of a coin") to start with one of the two pretzel groups (wheat or soy pretzel with safflower oil) for your first treatment period and then switch to the other safflower oil pretzel at your second treatment period.

DETAILED DESCRIPTION:
The overarching goal is to develop new dietary strategies to help postmenopausal women maintain a healthy weight by improving the availability of nutritious snacks that contain added health benefits and will be used to assess the impact of a functional snack on snacking behavior. The primary objective is to evaluate safflower oil delivered in a wheat pretzel compared to a wheat pretzel enhanced with soy will have a greater affect on blood triglyceride and glucose levels thereby affecting satiety and snacking behavior. The investigators hypothesize that a functional snack food such as a soft pretzel containing safflower oil either with or without soy compared to the control pretzel (wheat pretzel with no safflower oil) will reduce postprandial blood triglycerides and glucose.

This proposed multidisciplinary study is a randomized cross-over trial involving 20 overweight (BMI > 25 kg/m2) postmenopausal women with metabolic syndrome will participate in a dietary intervention study for a total of 14 weeks (two weeks of washout and three 4 week interventions). The study will require five visits to the Ohio State University Clinical Research Center (CRC), part of the Center for Clinical and Translational Sciences, Figure 5. Women will visit the CRC to be screened (Day-14) and their eligibility will be determined using a health and lifestyle questionnaire and results from a 12 hour fasting lipid panel (total cholesterol, LDL, HDL, triglycerides). Those meeting the National Cholesterol Education Program criteria for metabolic syndrome and having no other excluding conditions will be enrolled. Prior to their oral triglyceride tolerance tests (OTTT), women will be instructed to abstain from a. alcohol consumption for 72 hour, b. consume ≥150g of carbohydrates for 24 hours, c. abstain from vigorous exercise for 24 hours, d. collect urine for 24 hours, e. fast for 12 hours prior to all their clinic visits. When women arrive at the CRC for their clinic visits, weight and vital signs will be collected and a venous catheter placed for timed blood collections. Blood will be collected for serum triglycerides and glucose prior to (-5 minutes) and at 30, 60, 90, 120, 150, 180, 240, 300, and 360 minutes after consumption of the test meal. At their run-in visit (Day 0), subjects will consume a control pretzel with a flavored oil dip containing a standardized quantity of triglycerides (50 g long chain fatty acids). At the first treatment period (Day 28) visit, women will be randomized to one of the two intervention groups (wheat or soy pretzel with safflower oil) and then crossover to the other safflower oil pretzel at their second treatment period visit (Day 56). The two intervention pretzel meals will be accompanied with the same oil dip provided before. At the end of each OTTT visit women will be instructed to continue eating the test pretzels (12 pretzel bites/day) for the next 28 days as a snack. Subjects will be instructed to complete questions pertaining to their satiety during their 7 hour stay. Women will return for their last visit on Day 84 to submit all completed study materials (survey, dietary recall, and daily intake journal), completed 24 hour urine collection, and blood collection.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women 45 to 70 years of age
* Stated to be postmenopausal and has a cessation of menstruation for greater than 12 months
* Have a body mass index ≥25 kg/m2
* Must meet three of the five following criteria12

  1. Have a waist circumference greater than 35 inches
  2. Fasting serum triglycerides of greater than 150 mg/dL
  3. Fasting high density lipoprotein (HDL) less than 40 mg/dL
  4. Fasting blood glucose greater than 100 mg/dL
  5. Systolic blood pressure greater than 130 mm Hg or diastolic blood pressure greater than 85 mm Hg
* Agree to consume a standardized vitamin/mineral supplement and avoid other nutrition and alternative supplements for the duration of the study
* Agree to follow a legume free diet and to document any accidental consumption of restricted foods each day of the study

Exclusion Criteria:

* Have an active metabolic or digestive illness including malabsorptive disorders, renal insufficiency, hepatic insufficiency, or had recent (within the year) gastrointestinal surgery.
* Have a history or have active hormone related diseases of the pituitary, thyroid or pancreas that currently require supplemental hormonal administration thyroid hormones, adrenocorticotropic hormone (ACTH), growth hormone or other endocrine disorders requiring hormone or insulin administration
* Have an active or a recent history of any condition that causes altered immunity such as chronic inflammatory disease, autoimmune disorders, cancer, anemia, and blood dyscrasias
* Are on cholesterol lowering medications which include but not limited to statins, niacin (vitamin B3), bile-acid resins, fibric acid derivatives, or cholesterol absorption inhibitors.
* Have a known allergy or food intolerance to ingredients in study products (wheat, soy, or safflower oil)
* Are strict vegans (no consumption of animal, fish or egg products)
* Are heavy alcohol consumers (defined as an average consumption of greater than 14 drinks/week)
* Have a history of cancer or currently undergoing treatment for cancer
* Have been on an antibiotic regime lasting for more than one week in the last 6 months
* Are currently on another study for weight loss or trying to actively lose weight or recently (last 3 months) started medications for weight loss.

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2025-07 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants having Serious and Non-serious Adverse Events. | Up to 3 months
  Standardized qualitative and quantitative toxicity criteria (NIH) will be employed to evaluate safety and toxicity of daily safflower oil consumption.
Number of Participants with 80% Adherence to Safflower Oil Pretzels | Up to 3 months
  The daily consumption of safflower oil pretzels with and without soy will be assessed with a daily dietary intake journal as well as with measures of isoflavone and linoleic acid metabolites in urine and blood, respectively.

SECONDARY OUTCOMES:
Number of Participants with Improved Satiety Visual Analogue Scale (VAS) with Safflower Oil Pretzel Snacks Compared to Control Pretzels. | Up to 3 months
  The impact of safflower oil pretzels with and without soy on snacking behavior and satiety will be measured by comparing visual analogue scale surveys, food frequency questionnaires, and total energy intake extracted from 24 hour dietary recalls.
Area Under the Concentration-Time Curve for Serum Triglyceride and Glucose | Before test meal, 30, 60, 90, 120, 150, 180, 240, 300, and 360 minutes after the test meal on Days 0, 28, and 56
  Postprandial triglycerides and glucose following consumption of a single meal consisting of safflower oil pretzels with or without soy will be compared to a control pretzel having neither safflower oil nor soy.

OTHER OUTCOMES:
Identify Number of Participants with Changes in Blood Gene Expression from Day 0 Compared to Day 84. | Up to 3 months
  Impact of safflower oil consumption on gene expression profiles and biomarkers relevant to energy metabolism will be examined and correlated to their isoflavonoid metabolic profile.
Isoflavone Metabolite Profile Collected from Urine on Days 0, 28, 56, and 84 | Up to 3 months
  Women will be classified by their isoflavone metabolites in urine and correlated with biological effects of safflower oil pretzel intervention and gene expression

CONTACTS AND LOCATIONS:
Overall Officials: Yael Vodovotz, Ph.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center Clinical Research Center, Columbus, Ohio, United States